CLINICAL TRIAL: NCT02570945
Title: Randomized Controlled Trial of a Pharmacist-physician Intervention Model to Reduce High-risk Drug Use by Elderly Inpatients
Brief Title: Trial of a Pharmacist-physician Intervention Model to Reduce High-risk Drug Use by Hospitalised Elderly Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other)
Responsible Party: Principal Investigator, Benoit Cossette, Principal investigator, Centre de recherche du Centre hospitalier universitaire de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-965
Record Dates: First submitted 2015-09-25; First posted 2015-10-07 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Potentially Inappropriate Medication Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Pharmacist-physician medication review
  Interventions: Procedure: Pharmacist-physician intervention to reduce high-risk medication use by elderly inpatients
- Control (No Intervention)

INTERVENTIONS:
Procedure: Pharmacist-physician intervention to reduce high-risk medication use by elderly inpatients
  Arms: Intervention

SUMMARY:
The study population will consist of all elderly (65 and older) patients hospitalized at the Centre hospitalier universitaire de Sherbrooke. The patients who present a pharmacotherapeutic problem will be randomly allocated between intervention and control groups. Practically, the relevant data will be extracted from the Electronic Medical Record (EMR) on a daily basis and analysed by a Computerized Alert System (CAS) to identify pharmacotherapeutic problems. These problems will be analysed a pharmacist specialised in geriatrics to determine their clinical relevance and the modifications that can be made. Clinically relevant pharmacotherapeutic problems will be discussed by the pharmacist and treating physician to establish the changes needed to optimize drug therapy. A geriatrician will also be available to assist the pharmacist in his initial assessment for particularly complex cases. For control patients, a CAS analysis will be conducted to identify patients with a pharmacotherapeutic problem but there will not be a formal discussion amongst the health care providers (usual care) and the physicians of the control group will provide usual care to their patients. The investigators believe that it is ethical to provide usual care to the control group since the beneficial impact on patients outcomes of the investigators' intervention has not been demonstrated.

Pharmacotherapeutic problems were prioritized by the CHUS Elderly Adapted Care-medication committee and are based on the Beers criteria with an emphasis on drugs involved in the development of delirium. Selected pharmacotherapeutic problems are: 1) For patients 75 and older: i) taking a PIM; ii) concomitant use of 4 or more drugs from a list of drugs active at the CNS; iii) positive test for delirium with a PIM; 2) For patients 65 years and older: i) taking levodopa (Parkinson indicator) with a PIM; ii) taking cholinesterase inhibitor or memantine (indicators of dementia) with a PIM. The use of levodopa, a cholinesterase inhibitor or memantine are frailty indicators.

ELIGIBILITY:
Inclusion Criteria:

* Patients 65 and older admitted at the Centre hospitalier universitaire de Sherbrooke

Exclusion Criteria:

* Patients admitted in psychiatry and intensive care
* Patients seen only in the emergency room

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 321 (Actual)
Dates: Start 2015-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change rate in medication | 48 hours
  The main outcome was the change rate in medications, defined as the number of patient-days with a change in at least one medication out of the total number of patient-days with a pharmacist intervention with the treating physician.

SECONDARY OUTCOMES:
Clinical relevance of the Computerized Alert System alerts | 1 day
  The clinical relevance of the CAS alerts is defined as the proportion of alerts requiring an intervention (as assessed by the pharmacist) out of the total number of alerts.
Number of falls | From randomisation to the end of the hospitalisation, an average of 12 days
  Falls documented in the discharge summary and in the incident reports will be included
Delirium | From randomisation to the end of the hospitalisation, an average of 12 days
  Delirium will be assessed with the Confusion assessment Method (CAM) questionnaire
Death | From randomisation to the end of the hospitalisation, an average of 12 days
  Death
Readmission within 30 days of hospital discharge | 30 days after hospital discharge